CLINICAL TRIAL: NCT06384066
Title: Evaluation of a Mobile Health Application to Improve Patient Satisfaction and Outcomes After Urethroplasty: a Prospective Randomized Controlled Trial
Brief Title: Mobile Health Application to Improve Patient Satisfaction After Urethroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study team will not pursue this study moving forward. There have been no patients enrolled and the project will not continue. Study has been terminated with the IRB.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Ziho Lee, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00219774
Record Dates: First submitted 2024-02-19; First posted 2024-04-25 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Urethral Stricture
MeSH Terms: conditions — Urethral Stricture | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Other): Standard Care
  Interventions: Other: Standard of Care
- Standard Care + GetWell App (Other)
  Interventions: Other: GetWell Mobile Application; Other: Standard of Care

INTERVENTIONS:
Other: GetWell Mobile Application — GetWell utilizes an interactive health care application to allow patients to participate in their care. We plan to work with GetWell to develop a custom built plan for urethroplasty patients and provide patient education.
  Arms: Standard Care + GetWell App
Other: Standard of Care — Office Based Pathway

SUMMARY:
Create a custom urethroplasty mobile application that will guide patients through through the surgical process.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have a Urethral stricture and are under going urethroplasty surgery

Exclusion Criteria:

* Patients that do not have mobile phone capabilities
* Patients who have physical or cognitive impairment when using a mobile phone or answering questionnaires
* Inability to provide consent to the study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-28 (Estimated); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Improve patient satisfaction, education and reported outcomes | 0 to 3 months
  Asses through Patient reported outcome measurement survey, Urethral Stricture Symptom and Impact Measurement and Patient-Reported Outcomes Measurement information System 29-item profile (PROMIS) which assesses pain intensity using a 0-10 rating item, with higher scores being a worse outcome.
Change in rate of patient phone calls and messages | 0 to 12 months
  assess through chart review to evaluate the number of chart messages and phone calls
Rate of emergency department visits | 0 to 12 months
  Assess through chart review and patient reporting events.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT06384066/Prot_000.pdf